CLINICAL TRIAL: NCT06714669
Title: Comparison of General Anesthesia Hemodynamics Between Remimazolam and Propofol in Patients Undergoing Laparoscopic Hepatectomy: a Randomized, Controlled Trial.
Brief Title: Comparison of General Anesthesia Hemodynamics Between R and P in Patients Undergoing Laparoscopic Hepatectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongguo Zhou, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zhongguo Zhou
Record Dates: First submitted 2024-11-22; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Hypotension During Surgery
Keywords: hypotension; hemodynamics; general anesthesia; remimazolam; propofol
MeSH Terms: conditions — Hypotension | interventions — Propofol; remimazolam

STUDY DESIGN:
Intervention Model Description: participants in the experimental group used remimazolam as intravenous anesthetics while participants in the control group used propofol.
Who Masked: Participant, Care Provider
Masking Description: In order to ensure the management of perioperative anesthesia and the safety of patients, this study is a single-blind study, that is, anesthesiologists know what kind of anesthesia they have received, and carry out anesthesia plans for patients according to groups (group P / R). Participants and postoperative evaluators will not know the grouping of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm: Remimazolam Group (Experimental): Experimental Group (Remimazolam Anesthesia Arm): Patients in this arm will receive Remimazolam as the primary anesthetic agent for inducing and maintaining general anesthesia. The specific dosing regimen and administration protocol for Remimazolam will be determined based on the patient's characteristics and the surgical procedure being performed. Close monitoring of the patient's vital signs, particularly hemodynamic parameters, will be conducted throughout the anesthesia period to ensure safety and efficacy.
  Interventions: Drug: Remimazolam
- Control Arm: Propofol Group (Active Comparator): Control Group (Propofol Anesthesia Arm):
  Patients in this arm will receive Propofol as the primary anesthetic agent for general anesthesia. Propofol is a well-established anesthetic drug commonly used in clinical practice for its rapid onset and short duration of action. Similar to the experimental group, the dosing regimen and administration protocol for Propofol will be tailored to the individual patient's needs and the surgical procedure. Hemodynamic stability and other vital signs will also be closely monitored in this group to assess the safety and effectiveness of Propofol in comparison to Remimazolam.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — Control Group (Propofol Anesthesia Arm):
  Patients in this arm will receive Propofol as the primary anesthetic agent for general anesthesia. Propofol is a well-established anesthetic drug commonly used in clinical practice for its rapid onset and short duration of action. Similar to the experimental group, the dosing regimen and administration protocol for Propofol will be tailored to the individual patient's needs and the surgical procedure. Hemodynamic stability and other vital signs will also be closely monitored in this group to assess the safety and effectiveness of Propofol in comparison to Remimazolam.
  Arms: Control Arm: Propofol Group
Drug: Remimazolam — Experimental Group (Remimazolam Anesthesia Arm):
  Patients in this arm will receive Remimazolam as the primary anesthetic agent for inducing and maintaining general anesthesia. Remimazolam belongs to a new class of benzodiazepines and acts by enhancing the activity of GABAA receptors, leading to sedation and anesthesia. The specific dosing regimen and administration protocol for Remimazolam will be determined based on the patient's characteristics and the surgical procedure being performed. Close monitoring of the patient's vital signs, particularly hemodynamic parameters, will be conducted throughout the anesthesia period to ensure safety and efficacy.
  Arms: Experimental Arm: Remimazolam Group

SUMMARY:
This study is a randomized controlled trial designed to investigate the effects of two anesthetics, remimazolam and propofol, on intraoperative hemodynamics in patients undergoing laparoscopic liver resection. The experimental group receives remimazolam, while the control group receives propofol. The primary objective is to compare the hemodynamic responses of patients in both groups during the surgical procedure, aiming to provide insights into the potential differences in cardiovascular stability and anesthetic management associated with these two drugs

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for LMH;
* Age 18-80 years, BMI 18-28 kg/m2;
* American Association of Anesthesiologists（ASA）I-III;
* Child-Pugh grade A or B;
* No serious heart, brain and other important organ lesions;
* Informed and consent, and signed informed consent.

Exclusion Criteria:

* ASA IV-V or Child-Pugh C;
* Left ventricular ejection fraction (EF) <30%;
* Implanted with temporary or permanent pacemakers;
* Organic heart disease;
* Uncontrolled hypertension, diabetes and other chronic diseases;
* Prolonged use of sedative and analgesic drugs (such as opioid analgesics, benzodiazepines, antianxiety, antidepressants, antipsychotics, etc.);
* Alcohol addiction;
* Allergic to benzodiazepines or propofol, or to any ingredient in the studied drug;
* Known history of allergy to other anesthetics; difficulty in airway and intubation during induction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure | From enrollment to the end of treatment at 4 weeks
  The primary focus is to evaluate and compare the impact of Remimazolam and Propofol on hemodynamic parameters such as blood pressure (both systolic and diastolic). The objective is to assess whether Remimazolam causes less hemodynamic fluctuation compared to Propofol during the induction and maintenance of general anesthesia.
Heart rate | From enrollment to the end of treatment at 4 weeks
  The primary focus is to evaluate and compare the impact of Remimazolam and Propofol on hemodynamic parameters such as heart rate. The objective is to assess whether Remimazolam causes less hemodynamic fluctuation compared to Propofol during the induction and maintenance of general anesthesia.
Mean arterial pressure | From enrollment to the end of treatment at 4 weeks
  The primary focus is to evaluate and compare the impact of Remimazolam and Propofol on hemodynamic parameters such as mean arterial pressure. The objective is to assess whether Remimazolam causes less hemodynamic fluctuation compared to Propofol during the induction and maintenance of general anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-san University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No